CLINICAL TRIAL: NCT02127632
Title: Comparison of Laryngeal Mask Airway Supreme and Endotracheal Tube In Patients Undergoing Gynecological Laparoscopy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Sule Ozbilgin, Anaesthesiology and Reanimation, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 533-GOA
Record Dates: First submitted 2014-04-26; First posted 2014-05-01 (Estimated); Results first posted 2017-12-21 (Actual); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Anaesthesia
Keywords: laryngeal mask Supreme; laparoscopic gynecologic surgery; Laryngeal mask during surgery

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group ETT (endo tracheal tube) (Active Comparator): Group ETT (Endotracheal tube Group). In the ETT group for women no. 7-7.5 tube will use. ETT:Ruschelit, Teleflex Medical Snd. Bhd. Malaysia. Ref:112482
  Interventions: Device: Endotracheal Tube
- Group LM-S(Laryngeal mask supreme Group) (Experimental): Experimental: Group LM-S Group LM-S (Laryngeal mask supreme Group) For <50 kg, no. 3 Between 50-70 kg, no. 4 Between 70-100 kg, no. 5 LM-S (The Laryngeal Mask Company Limited, Singapore) will insert.
  Interventions: Device: Laryngeal Mask Airway-Supreme

INTERVENTIONS:
Device: Endotracheal Tube — ETT:Ruschelit, Teleflex Medical Snd. Bhd. Malaysia. Ref:112482
  Other Names: Device: Endotracheal Tube (ETT)
  Arms: Group ETT (endo tracheal tube)
Device: Laryngeal Mask Airway-Supreme — Before LM-S was inserted, to lubricate the surface in contact with the palate a water-based K-YTM gel (Johnson & Johnson Ltd. Maidenhead, UK) without local anesthetic was applied to completely cover the LM-S cuff. Depending on the patient's body weight For <50 kg, no. 3 Between 50-70 kg, no. 4 Between 70-100 kg, no. 5 LM-S (The Laryngeal Mask Company Limited, Singapore) was inserted.
  Other Names:
  LM-S (The Laryngeal Mask Company Limited, Singapore) serial number: 175030 lot: hmabw7
  Other Names: Group LM-S (laryngeal mask group).
  Arms: Group LM-S(Laryngeal mask supreme Group)

SUMMARY:
Endotracheal Tube (ETT) is still preferred for laparoscopic surgeries because of the fear of pulmonary aspiration and inadequate ventilation. Laryngeal mask Supreme (LM-S) is a single use device and the presence of a drain tube allows to separate the gastrointestinal and respiratory tracts. We planned to compare ventilation parameters and gastric distension scores of with LM-S vs ETT during laparoscopic gynecological surgery.

DETAILED DESCRIPTION:
This prospective, randomized and double-blind study received permission from "Dokuz Eylül University Medical Faculty Non-Interventional Research Ethics Committee" and after obtaining patients' informed consent, 100 patients with American society of anesthesiologists (ASA) classification group I-II, between 18-65 years, undergoing elective laparoscopic gynecological surgery were included.

Patients were divided into:

Group 1=>ETT (Endo tracheal group) (50 patients) Group 2=>LM-S (Laryngeal mask Supreme) (50 patients) Patients and surgeons performing the operation were not aware of which airway device was used. The patients in the groups were determined by block randomized methods.

Patients taken to the surgical room were given standard monitoring (non-invasive blood pressure measurements, electrocardiogram, and peripheral oxygen saturation measurements) before anesthesia induction. For preoperative sedation 0.02 mg/kg midazolam IV was administered.

Patients were preoxygenated with 6 L/min oxygen for 3 minutes through a face mask.

For anesthesia induction after 2 minutes of 0.2 µg/kg/min remifentanil and 6 mg/kg/hr propofol infusion, IV 1-2 mg/kg propofol , 0,5 mg/kg rocuronium bromide was administered. After induction patients were ventilated with 6 L/min 100% oxygen through a face mask.

Airway devices were inserted by two researchers with more than 5 years experience.

Anesthetic maintenance was provided by 50% O2/air mixture with 0.1-0.4 µg/kg/min remifentanil and 50-150 µg/kg/hr (3-9 mg/kg/hr) propofol IV infusion (24).

Before LM-S was inserted, to lubricate the surface in contact with the palate a water-based gel without local anesthetic was applied to completely cover the LM-S cuff. Depending on the patient's body weight For <50 kg, no. 3 Between 50-70 kg, no. 4 Between 70-100 kg, no. 5 LM-S (The Laryngeal Mask Company Limited, Singapore) was inserted.

After LM-S placement the cuff was inflated with air so as to have a pressure below 60 water of centimeter (cmH20) (cuff pressure manometer, Rusch, Germany). Two minutes after LM-S placement, before insufflation, 10 minutes after insufflation and trendelenburg position, before desufflation and before LM-S removal, cuff pressure was measured repeatedly and recorded. At the same time intervals in the ETT group, ETT cuff pressure was measured.

In the ETT group for women no. 7-7.5 tube was used. The ETT cuff was inflated until the leak sound ceased. It was measured with a manometer to remain between 20-30 water of centimeter (cmH20).

Successful placement of LM-S or ETT was confirmed by square-shaped waves observed on the capnogram, easy ventilation of the respiration balloon and visible chest movements. After successful placement of the airway device, it was covered to prevent observation of which device was used.

The length of time for successful placement (duration from mouth opening to first successful ventilation), number of tries, and ease of placement were recorded. Ease of placement was evaluated by the anesthetist in charge of the airway as easy, hard or unsuccessful (alternative airway management).

In a situation where airway provision was unsuccessful after 3 tries, patients without placement of LM-S or who could not be intubated were switched to the other group and airway management was provided.

For oropharyngeal leak test after the expiratory valve was closed air was shut off, O2 was reduced to 3 L/min and the first pressure value when a leak sound was heard was recorded as the oropharyngeal leak pressure. To prevent exposure of the lungs to barotrauma, when the peak inspiratory pressure reached 40 cmH2O the expiratory valve was opened and the test was concluded. This test was repeated before peritoneal insufflation, 10 minutes later and immediately before desufflation and was completed by a researcher blind to the type of airway device inserted.

Positive pressure respiration was begun by using a ring system, 2-4 L/min fresh gas flow and 0.5 fraction of inspired oxygen (FiO2) volume controlled 6-8 ml/kg tidal volume and 10 respirations/min frequency. PEEP was not administered and I:E ratio was adjusted to 1:2. ETCO2 was held between 35-45 mmHg, if necessary first respiration frequency was increased then tidal volume was increased. Permission was given for CO2 insufflation for the laparoscopic intervention with peritoneal interior pressure of 15 mmHg.

Two minutes after LM-S or ETT placement, before insufflation, 10 minutes after insufflation and trendelenburg position, immediately before peritoneal desufflation and before airway device removal, ventilation parameters were evaluated.

Respiratory measurements to be recorded: Tidal volume (TV), respiration number (RN), peripheral oxygen saturation (SPO2), end-tidal carbon dioxide pressure (PETCO2), peak airway pressure (P peak), mean airway pressure (P mean) and expiration volume per minute (VE).

Hemodynamic measurements to be recorded: (simultaneous to the measurements above and additionally before induction) Systolic blood pressure (SBP), diastolic blood pressure (DBP), mean blood pressure (MBP) and heart rate (HR).

Evaluation related to gastric tube:

Immediately after airway device placement using either the LM-S drainage tube or in intubated patients using a 14 Ch orogastric probe within the airway, the stomach was reached and the gastric contents were aspirated. Ease of placement and amount of fluids aspirated were recorded. Ease of placement was classified by the person who inserted the orogastric probe as very easy, easy, difficult and very difficult.

Immediately after the intra-abdominal laparoscopic intervention and immediately before peritoneal insufflation was ended, gastric distension was evaluated by a surgeon blind to the airway device used between 0-10 (0=empty stomach, 10=distension obstructing the surgical field) and the difference between the scores at the start and end of the operation was recorded .

When the patient cooperated LM-S or ETT was removed and total anesthesia duration and peritoneal insufflation duration was recorded. Possible complications that could develop during airway device removal (coughing, vomiting, laryngeal stridor, laryngeal spasm or requirement for airway intervention) were recorded.

After LM-S removal the presence of blood was evaluated as

1. no blood
2. trace amounts of blood
3. clear amount of blood Revived patients were taken to the recovery unit and a blind researcher evaluated the patients' throat pain, hoarseness and presence of difficulty swallowing in the 1st and 24th hours. To evaluate throat pain the visual analogue scale was used.

ELIGIBILITY:
Inclusion Criteria:

* ASA classification group I-II
* Between 18-65 years
* Undergoing elective laparoscopic gynecological surgery

Exclusion Criteria:

* Individuals with any neck and upper respiratory pathology
* Individuals at risk of gastric content regurgitation/aspiration (previous upper gastrointestinal surgery, known hiatus hernia, gastroesophageal reflux, history of peptic ulcer, full stomach, pregnancy)
* Individuals with low pulmonary compliance or high airway resistance (chronic lung diseases)
* Obese patients (BMI >35)
* Individuals with sore throat, dysphagia and dysphonia
* Individuals with possibility or history of difficult airway
* Operation time planned for more than 4 hours

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: BAHAR KUVAKİ, M.D., Principal Investigator — Dokuz Eylül University, School of Medicine, Department of Anesthesiology and Reanimation
Locations (1):
- Sule Ozbilgin, Izmi̇r, Narlıdere, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kuvaki B, Ozbilgin S, Gunenc SF, Kucuk BA. Comparison of LM-Supreme and endotracheal tube in patients undergoing gynecological laparoscopic surgery. J Clin Monit Comput. 2020 Apr;34(2):295-301. doi: 10.1007/s10877-019-00310-2. Epub 2019 Apr 9. PMID 30968326

RESULTS

PARTICIPANT FLOW:
Groups:
- Group ETT (Endo Tracheal Tube): Group ETT (Endotracheal tube Group). In the ETT group for women no. 7-7.5 tube will use. ETT:Ruschelit, Teleflex Medical Snd. Bhd. Malaysia. Ref:112482
  Laryngeal Mask Airway-Supreme: Before LM-S was inserted, to lubricate the surface in contact with the palate a water-based gel without local anesthetic was applied to completely cover the LM-S cuff. Depending on the patient's body weight For <50 kg, no. 3 Between 50-70 kg, no. 4 Between 70-100 kg, no. 5 LM-S (The Laryngeal Mask Company Limited, Singapore) was inserted.
  Other Names:
  LM-S (The Laryngeal Mask Company Limited, Singapore) serial number: 175030 lot: hmabw7
- Group LM-S(Laryngeal Mask Supreme Group): Experimental: Group LM-S Group LM-S (Laryngeal mask supreme Group) For <50 kg, no. 3 Between 50-70 kg, no. 4 Between 70-100 kg, no. 5 LM-S (The Laryngeal Mask Company Limited, Singapore) will insert.
  Endotracheal Tube: ETT:Ruschelit, Teleflex Medical Snd. Bhd. Malaysia. Ref:112482
Period: Overall Study
Arm/Group | Group ETT (Endo Tracheal Tube) | Group LM-S(Laryngeal Mask Supreme Group)
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group ETT (Endo Tracheal Tube): Group ETT (Endotracheal tube Group). In the ETT group for women no. 7-7.5 tube will use. ETT:Ruschelit, Teleflex Medical Snd. Bhd. Malaysia. Ref:112482
  Laryngeal Mask Airway-Supreme: Before LM-S was inserted, to lubricate the surface in contact with the palate a water-based K-YTM gel (Johnson & Johnson Ltd. Maidenhead, UK) without local anesthetic was applied to completely cover the LM-S cuff. Depending on the patient's body weight For <50 kg, no. 3 Between 50-70 kg, no. 4 Between 70-100 kg, no. 5 LM-S (The Laryngeal Mask Company Limited, Singapore) was inserted.
  Other Names:
  LM-S (The Laryngeal Mask Company Limited, Singapore) serial number: 175030 lot: hmabw7
- Total: Total of all reporting groups
Arm/Group | Group ETT (Endo Tracheal Tube) | Group LM-S(Laryngeal Mask Supreme Group) | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.36 (11.52) | 38.86 (11.48) | 39.11 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Mean Airway Pressures
Description: The measure is the mean airway pressure (cmH2O):
  T1= 2 minutes after airway device insertion T2= 10 minutes after insufflation T3= Before desufflation T4= Before removal of airway device
Time Frame: At first and last 10 minutes of pneumoperitoneum
Measure: Mean (Full Range); unit: cmH20
Arm/Group | Group ETT (Endo Tracheal Tube) | Group LM-S(Laryngeal Mask Supreme Group)
Number analyzed (Participants) | 50 | 50
cmH20
  T1 | 7 [5 to 9] | 6 [4 to 9]
  T2 | 8 [6 to 12] | 8 [6 to 19]
  T3 | 8 [6 to 12] | 8 [4 to 17]
  T4 | 7 [5 to 11] | 7 [5 to 12]

2. Secondary Outcome: Evaluation of Gastric Distention
Description: To provide the adequate gastric distention of either the LM-Supreme or the tracheal tube, as assigned. Gastric distension was evaluated by a surgeon blind to the airway device used between 0-10 (0=empty stomach, 10=distension obstructing the surgical field)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group ETT (Endo Tracheal Tube) | Group LM-S(Laryngeal Mask Supreme Group)
Number analyzed (Participants) | 50 | 50
units on a scale | 3.24 (1.99) | 2.02 (1.07)

3. Secondary Outcome: Throat Pain According to Visual Analogue Scale
Description: Patients were asked about the presence of sore throat - defined as the presence of constant pain in the throat, 1 hr and 24 hr after the end of surgery according to Visual Analogue Scale. (range min. 0, max.10; >4 analgesia planned)
Time Frame: postoperative 1st and 24th hours
Measure: Mean (Standard Deviation); unit: point
Arm/Group | Group ETT (Endo Tracheal Tube) | Group LM-S(Laryngeal Mask Supreme Group)
Number analyzed (Participants) | 50 | 50
point
  postoperative 1st hour | 2.04 (1.61) | 0.32 (0.76)
  postoperative 24th hours | 0 (0) | 0 (0)

ADVERSE EVENTS:
Arm/Group | Group ETT (Endo Tracheal Tube) | Group LM-S(Laryngeal Mask Supreme Group)
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

LIMITATIONS AND CAVEATS:
We studied a female population with normal airways undergoing elective gynaecological laparoscopic surgery.

Second, we only studied non-obese patients. Third we excluded cases with difficult airway.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No